CLINICAL TRIAL: NCT03475342
Title: Tranexamic Acid for the Prevention of Postpartum Bleeding in Women With Anaemia: an International, Randomised, Double-blind, Placebo Controlled Trial.
Brief Title: World Maternal Antifibrinolytic Trial_2
Acronym: WOMAN-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Wellcome Trust (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WOMAN_2; 03475342 (Other: ISRCTN)
Record Dates: First submitted 2018-02-23; First posted 2018-03-23 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-04

CONDITIONS: Intrapartum - Moderate and Severe Anaemia
Keywords: prevention, postpartum haemorrhage; moderate anaemia; severe anaemia; antifibrinolytic; tranexamic acid; pregnancy; pain; episiotomy
MeSH Terms: conditions — Anemia; Postpartum Hemorrhage; Pain | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A randomised, double blind, placebo controlled trial among 15,000 women with moderate or severe anaemia having given birth vaginally.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking was done by an independent clinical trials supply company. It will involve the removal of the original manufacturer's label and replacement with the clinical trial label bearing the randomisation number, which will be used as the pack identification. Apart from the randomisation number, all pack label texts will be identical for tranexamic acid and placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Active Comparator): One intravenous injection of tranexamic acid. Total dose 1 gram (10mL)
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): One Injection of the placebo which is 10 mL Sodium Chloride (0.9%)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid — Ampoules and packaging for both arms will be identical in appearance.
  Arms: Tranexamic acid
Other: Placebo — Ampoules and packaging for both arms will be identical in appearance.
  Other Names: (Sodium Chloride 0.9%)
  Arms: Placebo

SUMMARY:
Postpartum haemorrhage (PPH) is responsible for about 100,000 maternal deaths every year, almost all of which occur in low and middle income countries. When given within three hours of birth, tranexamic acid reduces deaths due to bleeding in women with PPH by almost one third. However, for many women, treatment of PPH is too late to prevent death and severe morbidities. Over one-third of pregnant women in the world are anaemic and many are severely anaemic. We now want to do the WOMAN-2 trial to see if giving tranexamic acid can prevent PPH and other severe outcomes in women with moderate and severe anaemia.

DETAILED DESCRIPTION:
Anaemia is a cause and consequence of PPH. A cohort study in Assam, India found that women with moderate or severe anaemia had a greatly increased risk of PPH. Women with moderate anaemia had a 50% increased risk, whereas those with severe anaemia had a ten-fold increased risk of PPH. Anaemic women may be more susceptible to uterine atony due to impaired oxygen transport to the uterus. Anaemic women experience worse outcomes after PPH. An international survey of 275,000 women found that severe maternal outcomes after PPH were nearly three times more common in anaemic than in non-anaemic women. Even moderate bleeding can be life threatening in anaemic women. Excessive bleeding after childbirth worsens maternal anaemia, resulting in a vicious circle of bleeding and adverse outcomes. Fatigue due to anaemia severely limits a mothers' wellbeing and her ability to care for her children. Despite efforts to prevent anaemia, many women labour with perilously low haemoglobin levels

Tranexamic acid (TXA) inhibits fibrinolysis by blocking the lysine binding sites on plasminogen. TXA reduces surgical bleeding and death due to bleeding in trauma patients. The WOMAN trial assessed the effects of TXA in 20,060 women with PPH. When given within three hours of birth, TXA reduced death due to bleeding by nearly one-third (RR=0.69, 95% CI 0.52 to 0.91, p=0.008). However, for many women, treatment is too late to prevent death from PPH. Most PPH deaths occur in the first hours after giving birth and women with anaemia are at greatly increased risk. Whilst there have been some trials of TXA for the prevention of PPH, most have serious flaws and none collected data on maternal health and wellbeing. There is currently no reliable evidence about the effectiveness and safety of TXA for preventing PPH.

The WOMAN-2 trial will determine reliably the effects of TXA in anaemic women who give birth vaginally.

We will also conduct a pre-planned cohort analysis of data from the WOMAN-2 trial to assess the effect of pain control and episiotomy on the risk of post-partum haemorrhage. Adrenaline is a potent stimulus for fibrinolysis. Adrenaline causes the release of tissue plasminogen activator (TPA) from the endothelium. In trauma victims, high adrenaline levels are associated with increased fibrinolysis, decreased clot strength and increased deaths due to bleeding. Childbirth is intensely painful and maternal adrenaline levels are two to six times higher during labour. Maternal adrenaline concentrations peak in the second and third stages of labour but then rapidly return to normal after birth. Pain control can reduce the maternal catecholamine response. We hypothesize that painful procedures such as episiotomy will significantly increase the risk of postpartum haemorrhage and that pain control will reduce the risk of PPH.

The exposures of interest are the presence or absence of pain control during labour and delivery and whether episiotomy was conducted prior to birth. Pain control will be categorised as present or absent but the type of pain control administered during labour will also be described and examined. The types of pain control recorded in the study are epidural, opioids, 'other', or a combination of opioids and other pain control. For the multivariable regression analysis, the pain control variable was converted into a binary variable indicating whether a participant received any pain control or not. Episiotomy will be categorised as present or absent according to the CRF. The main outcome variable will be a clinical diagnosis of PPH (binary: yes/no), defined as an estimated blood loss of more than 500 mL or any blood loss sufficient to compromise haemodynamic stability within 24 hours. Potential confounding factors will include maternal age, BMI, anaemia, history of PPH, antepartum hemorrhage, hypertensive disease, multiple gestation, parity, prophylactic uterotonics, duration of labor, induction and augmentation of labor, assisted delivery, gestational age, birth canal trauma, placental abruption, and macrosomia.

We will use multivariable logistic regression to examine the association between pain control and episiotomy and the risk of PPH after adjusting for confounding factors. We will describe our causal assumptions using a directed acyclic graph. We will examine the association between the exposures of interest and PPH with odds ratios and 95% confidence intervals. We will estimate odds ratios and 95% CI for the crude association between the exposures of interest and PPH and after controlling for confounding factors. We will check for collinearity using variance inflation factors. Finally, we will examine whether the effect of pain control and episiotomy on the risk of PPH is modified by tranexamic acid treatment. To do this we will conduct stratified analysis and calculate a p-value for heterogeneity using a likelihood ratio test.

ELIGIBILITY:
Inclusion Criteria:

* Women with moderate or severe anaemia (haemoglobin level <100 g/L or packed cell volume <30%) after giving birth vaginally where the responsible clinician is substantially uncertain whether to use TXA

Exclusion Criteria:

* Women who are not legally adult (<18 years) and not accompanied by a guardian
* Women with a known allergy to tranexamic acid or its excipients
* Women who experience postpartum haemorrhage before the umbilical cord is cut or clamped.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women who have given birth
Enrollment: 15068 (Actual)
Dates: Start 2019-08-24 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-10-29 (Actual)

PRIMARY OUTCOMES:
Postpartum Haemorrhage (cause will be described) | 24 hours after administration of the trial medication or at discharge from hospital, whichever is earlier
  Clinical assessment: This may be an estimated blood loss of more than 500 mL or any blood loss sufficient to compromise haemodynamic stability within 24 hours of delivery. Haemodynamic instability is based on clinical judgement and assessed using clinical signs (low systolic blood pressure, tachycardia, reduced urine output).

SECONDARY OUTCOMES:
Postpartum blood loss | 24 hours after administration of the trial medication or at discharge from hospital, whichever is earlier
  Clinical assessment
Haemoglobin | 24 hours after administration of the trial medication or at discharge from hospital, whichever is earlier
  Haemocue (Point of care test)
Haemodynamic instability | 24 hours after administration of trial treatment or discharge from hospital, whichever is earlier
  Defined as per protocol
Shock index | 24 hours after administration of trial treatment or discharge from hospital, whichever is earlier
  Heart rate/systolic blood pressure
Quality of Life (maternal) | Day 42 or discharge from hospital, whichever is earlier
  Defined as per protocol
Expected side effects of trial medication | Day 42 or discharge from hospital, whichever is earlier
  nausea, vomiting, diarrhoea
Exercise tolerance | Day 42 or discharge from hospital, whichever is earlier
  6 minute walk test
Interventions to control primary postpartum haemorrhage (medical and surgical) | Day 42 or discharge from hospital, whichever is earlier
  Any of the following: uterotonics, removal of placenta/placenta fragments, intrauterine balloon tamponade, bimanual uterine compression, external aortic compression, non-pneumatic anti-shock garments, uterine artery embolisation, uterine compression suture, hysterectomy and laparotomy to control bleeding
Receipt of blood product transfusion | Day 42 or discharge of mother from hospital, whichever is earlier
  units and type
Vascular occlusive events | Day 42 or discharge from hospital, whichever is earlier
  Any of the following:pulmonary embolism (PE), deep vein thrombosis (DVT), stroke, myocardial infarction
Symptoms of anaemia | Day 42 or discharge of mother from hospital, whichever is earlier
  measured using Quality of life Questionnaire and walk test
Organ disfunction | Day 42 or discharge from hospital, whichever is earlier
  Any of the following: Cardiovascular, Respiratory, Renal, Hepatic, Neurological, Coagulation/ haematologic dysfunction
Sepsis | Day 42 or discharge from hospital, whichever is earlier
  diagnosis is based on the presence of both infection and a systemic inflammatory response syndrome (SIRS). SIRS requires two or more of the following: a) temperature <36°C or >38°C (b) heart rate >90 beats/min (c) respiratory rate >20 breaths/min (d) white blood cell count <4x109/L (<4000/mm³) or >12x109/L (>12,000/mm³)
In hospital death | Day 42
  Cause and time of death will be described
Length of hospital stay. | Day 42 or discharge from hospital, whichever is earlier
  Days
Admission to and time spent in higher level facility | Day 42 or discharge from hospital, whichever is earlier
  High Dependency and/or Intensive Care Units
Status of baby/ies | Day 42 or discharge of mother from hospital, whichever is earlier
  alive or dead
Thromboembolic events in breastfed babies | Day 42 or discharge of mother from hospital, whichever is earlier
  as defined in protocol
Adverse events | Day 42
  Any untoward medical occurrence (other than expected complications)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Roberts, Study Chair — Clinical Trials Unit, London School of Hygiene and Tropical Medicine; Haleema Shakur-Still, Study Chair — Clinical Trials Unit, London School of Hygiene and Tropical Medicine; Rizwana Chaudhri, Principal Investigator — National Coordinating Investigator, Shifa Tameer-e-Millat University, Pakistan; Folasade A Bello, Principal Investigator — National Coordinating Investigator, College of Medicine, University of Ibadan, Nigeria; Bellington Vwalika, Principal Investigator — National Coordinating Investigator, University of Zambia School of Medicine, Zambia; Projestine Muganyizi, Principal Investigator — National Coordinating Investigator, Muhimbili University of Health and Allied Sciences, Tanzania; Oladapo Olayemi, Principal Investigator — National Coordinating Investigator, College of Medicine, University of Ibadan, Nigeria
Locations (41):
- Nigeria (7):
  - Mother & Child Hospital, Akure
  - University of Medical Sciences Teaching Hospital, Akure
  - Adeoyo Maternity Hospital, Ibadan
  - Ilorin General Hospital, Ilorin
  - Muhammad Abdullahi Wase Specialist Hospital, Kano
  - Ladoke Akintola University of Technology Teaching Hospital, Ogbomoso
  - State Hospital, Oyo
- Pakistan (25):
  - Ayub Teaching Hospital (Unit A), Abbottabad
  - Ayub Teaching Hospital (Unit C), Abbottabad
  - Ayub Teaching Hospital Unit B, Abbottabad
  - Bahawalpur Victoria Hospital, Bahawalpur
  - Aziz Bhatti Teaching Hospital, Gujrat
  - MCH PIMS, Islamabad
  - Military Hospital, Islamabad
  - Civil Hospital, Karachi
  - Jinnah Postgraduate Medical Centre, Karachi
  - Koohi Goth Hospital, Karachi
  - Jinnah Hospital, Lahore
  - Services Hospital, Lahore
  - Sir Ganga Ram Hospital Unit 1, Lahore
  - Sir Ganga Ram Hospital Unit 2, Lahore
  - Sir Ganga Ram Hospital Unit 3, Lahore
  - Sir Ganga Ram Hospital Unit 4, Lahore
  - Chandka SMBBMU Sheikh Zaid Woman Hospital Unit 1, Larkana
  - Chandka SMBBMU Sheikh Zaid Woman Hospital Units 2 & 3, Lārkāna
  - Nishtar Hospital Unit 1, Multan
  - Nishtar Hospital Unit 2, Multan Khurd
  - Nishtar Hospital Unit 3, Multan Khurd
  - Bolan Medical Centre, Quetta
  - Benazir Bhutto Shaheed Hospital, Rawalpindi
  - Federal Government Polyclinic, Rawalpindi
  - Holy Family Hospital, Rawalpindi
- Tanzania (8):
  - Mount Meru Regional Referral Hospital, Arusha
  - Amana Regional Referral Hospital,, Dar es Salaam
  - Muhimbili National Hospital, Dar es Salaam
  - Temeke Regional Referral Hospital, Dar es Salaam
  - Dodoma Regional Referral Hospital, Dodoma
  - Tumbi Regional Referral Hospital, Kibaha, Kibaha
  - Mwananyamala Regional Referral Hospital, Kinondoni
  - Mbeya Zonal Referral Hospital, Mbeya
- Women and Newborn Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared publicly when all planned analyses are completed by the Woman-2 Trial Collaborators. This will be hosted on freebird.lshtm.ac.uk
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared publicly when all planned analyses are completed by the Woman-2 Trial Collaborators.
Access Criteria: Totally anonymised data (without random allocation, patient, country and site identifiers) will be freely available.
  Where random allocation codes, country/site identifiers are requested, appropriate pre-specified analysis plan will need to be submitted to the Trial Management Group for review and if necessary, appropriate Ethics Committee approval will be required.
URL: http://freebird.lshtm.ac.uk

REFERENCES:
- [Derived] WOMAN-2 Trial Collaborators. The effect of tranexamic acid on postpartum bleeding in women with moderate and severe anaemia (WOMAN-2): an international, randomised, double-blind, placebo-controlled trial. Lancet. 2024 Oct 26;404(10463):1645-1656. doi: 10.1016/S0140-6736(24)01749-5. PMID 39461792
- [Derived] Larson NJ, Mergoum AM, Dries DJ, Cook A, Blondeau B, Rogers FB. THE ROLE OF TRANEXAMIC ACID IN POSTPARTUM HEMORRHAGE: A NARRATIVE REVIEW. Shock. 2024 Nov 1;62(5):620-627. doi: 10.1097/SHK.0000000000002455. Epub 2024 Aug 20. PMID 39162220
- [Derived] Collier T, Shakur-Still H, Roberts I, Balogun E, Olayemi O, Bello FA, Chaudhri R, Muganyizi P; WOMAN-2 Trial Collaborators. Tranexamic acid for the prevention of postpartum bleeding in women with anaemia: Statistical analysis plan for the WOMAN-2 trial: an international, randomised, placebo-controlled trial. Gates Open Res. 2023 Aug 3;7:69. doi: 10.12688/gatesopenres.14529.2. eCollection 2023. PMID 37664793
- [Derived] Brenner A, Roberts I, Balogun E, Bello FA, Chaudhri R, Fleming C, Javaid K, Kayani A, Lubeya MK, Mansukhani R, Olayemi O, Prowse D, Vwalika B, Shakur-Still H. Postpartum haemorrhage in anaemic women: assessing outcome measures for clinical trials. Trials. 2022 Mar 18;23(1):220. doi: 10.1186/s13063-022-06140-z. PMID 35303924
- [Derived] Ker K, Roberts I, Chaudhri R, Fawole B, Beaumont D, Balogun E, Prowse D, Pepple T, Javaid K, Kayani A, Arulkumaran S, Bates I, Shakur-Still H; WOMAN-2 trial collaborators. Tranexamic acid for the prevention of postpartum bleeding in women with anaemia: study protocol for an international, randomised, double-blind, placebo-controlled trial. Trials. 2018 Dec 29;19(1):712. doi: 10.1186/s13063-018-3081-x. PMID 30594227